CLINICAL TRIAL: NCT05835336
Title: A Pilot Study to Assess the Efficacy and Safety of a Novel Device (VIZO Glasses) in the Management of ADHD in Adolescents.
Brief Title: A Novel, Non-pharmacological, Intervention for the Management of ADHD in Adolescents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VIZO Specs Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VIZO_004
Record Dates: First submitted 2023-04-18; First posted 2023-04-28 (Actual); Results first posted 2025-03-07 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2025-03

CONDITIONS: ADHD
Keywords: ADHD; Peripheral Retinal Stimulation; Non-pharmacological treatment; Adolescents
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Active (Experimental): VIZO Glasses- personalized
  Interventions: Device: VIZO Glasses

INTERVENTIONS:
Device: VIZO Glasses — Eyeglasses with personalized peripheral retinal stimuli

SUMMARY:
This is a 2-month study in which eligible ADHD adolescents will be provided with personalized VIZO Glasses

DETAILED DESCRIPTION:
This is a pilot, open-label study of a 2-month treatment with VIZO Glasses. Following the enrollment, the participants will go through an adjustment process where they will be fitted with a personalized pair of VIZO Glasses. The participants will be instructed to wear the glasses throughout the day for two months. A follow-up visit at the end of the 2-month treatment will be conducted to assess the efficacy of VIZO Glasses on managing ADHD symptoms, using the ADHD Rating Scale (ADHD-RS) parent-report questionnaire, the Behavior Rating Inventory of Executive Function (BRIEF), the Conners Continuous Performance Test-3, and the Clinical Global Impression-Improvement (CGI-I). Safety will be monitored by documentation of adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Documented history of primary ADHD diagnosis by certified clinicians
* Age 12-17 y
* Minimum total of 24 on the parent ADHD-IV Rating Scale (ADHD-RS)
* Written informed consent
* Able and willing to complete all required ratings and assessments

Exclusion Criteria:

* Any current psychiatric/neurological comorbidity (e.g., epilepsy, Autism, depression, TBI, etc.), other than ADHD
* ADHD Medications (stimulants, non-stimulants, other)
* Undergoing Neurofeedback, cognitive training

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 32 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2023-07-06 (Actual); Study Completion 2023-07-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Zohar Elyoseph, PhD, Principal Investigator — Max Stern Academic College of Emek Yezreel
Locations (1):
- Max Stern Academic College of Emek Yezreel, Haifa, Israel

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Thirty-two participants met the inclusion criteria. Three participants failed to complete the personalization process, resulting in 29 participants receiving the intervention.
Period: Overall Study
Arm/Group | Active
Started | 32
Received Intervention | 29 (Three participants did not complete the personalization process, and therefore did not receive the intervention.)
Completed | 24
Not Completed | 8
Not completed — Withdrawal by Subject | 5
Not completed — Did not complete the personalization process | 3

BASELINE CHARACTERISTICS:
Population: One participant excluded from per-protocol analysis due to a major protocol deviation.
Arm/Group | Active
Number analyzed (Participants) | 23
Age, Continuous [Mean (Standard Deviation); unit: years] | 14.67 (1.87)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 14
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
ADHD Rating Scale (ADHD-RS) Parent-report Questionnaire - Total Score [Mean (Standard Deviation); unit: units on a scale] | 30.30 (5.47)

OUTCOME MEASURES:

1. Primary Outcome: Change in the ADHD Rating Scale (ADHD-RS) Parent-report Questionnaire - Total Score - at Baseline and 2 Months Follow up
Description: The ADHD-RS is a parent report questionnaire that is used to aid in the diagnosis of ADHD in children ranging from ages 5-17. The questionnaire contains 18 symptom items corresponding to the DSM-V criteria for ADHD. The parent rates each symptom item on a 4-point Likert scale ranging from 0 ('Never or Rarely') to 3 ('Very Often'). The total score goes from 0 up to 54. Higher scores mean more symptoms and higher ADHD impairments.
Time Frame: Baseline, 2-month
Population: Three participants did not complete the questionnaire.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Active
Number analyzed (Participants) | 20
score on a scale
  Baseline | 30.30 (1.22)
  End of study | 22.85 (2.02)
Statistical Analysis 1: Comparison: Active; Test type: Superiority — Considering the exploratory nature of the study, a sample size of at least 0.5 (Cohen's D) for a 2-Tailed test, at alpha-0.05 with a power of 80%, was chosen to detect significant within-subject effects; p < 0.001, t-test, 2 sided; Mean Difference (Final Values) = 7.45

2. Primary Outcome: Change in the ADHD Rating Scale (ADHD-RS) Parent-report Questionnaire - Inattentiveness Subscale - at Baseline and 2 Months Follow up
Description: The Inattention subscale of the ADHD-RS contains 9 symptom items, that are designed to measure the child's attention level on tasks or play activities.The items are rated by the parent on a 4-point Likert scale ranging from 0 ('Never or Rarely') to 3 ('Very Often'). The total score goes from 0 up to 27. Higher scores mean more symptoms and higher ADHD impairments.
Time Frame: Baseline, 2-month
Population: Three participants did not complete the questionnaire.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Active
Number analyzed (Participants) | 20
score on a scale
  Baseline | 18.00 (0.93)
  End of study | 14.10 (1.16)
Statistical Analysis 1: Comparison: Active; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p < 0.001, t-test, 2 sided; Mean Difference (Final Values) = 3.9

3. Primary Outcome: Change in the ADHD Rating Scale (ADHD-RS) Parent-report Questionnaire - Hyperactivity-Impulsivity Subscale - at Baseline and 2 Months Follow up
Description: The Hyperactivity-Impulsivity subscale of the ADHD-RS contains 9 symptom items, that are designed to measure the child's hyperactivity level and impulsivity level. The items are rated by the parent on a 4-point Likert scale ranging from 0 ('Never or Rarely') to 3 ('Very Often'). The total score goes from 0 up to 27. Higher scores mean more symptoms and higher ADHD impairments.
Time Frame: Baseline, 2-month
Population: Three participants did not complete the questionnaire.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Active
Number analyzed (Participants) | 20
score on a scale
  Baseline | 12.30 (1.03)
  End of study | 8.75 (1.23)
Statistical Analysis 1: Comparison: Active; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.001, t-test, 2 sided; Mean Difference (Final Values) = 3.55

4. Primary Outcome: Change in Behavior Rating Inventory of Executive Function (BRIEF) - Metacognitive Index - at Baseline and 2 Months Follow up
Description: The Metacognition Index (MI) of the BRIEF reflects a child's ability to self-manage and monitor tasks cognitively. The subscale is composed of the Initiate, Working Memory, Plan/Organize, Organization of Materials, and Monitor scales of the BRIEF. It uses a Likert-type response format ranging from 1 to 3, where 1 is never, 2 is sometimes, and 3 is often. The MI subscale includes 40-items with score ranges between 0 to 120. Higher values represent worse outcome and greater difficulties with executive functions. High scores indicate executive deficit.
Time Frame: Baseline, 2-month
Population: Four participants did not complete the questionnaire.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Active
Number analyzed (Participants) | 19
score on a scale
  Baseline | 107.89 (2.11)
  End of study | 102.74 (2.94)
Statistical Analysis 1: Comparison: Active; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.032, t-test, 2 sided; Mean Difference (Final Values) = 5.16

5. Secondary Outcome: Clinical Global Impression-Improvement (CGI-I) - at 2 Months Follow up
Description: Based on an interview with the participant, the clinician rates the total improvement on a 7 point scale as follows: 1=very much improved since the initiation of treatment; 2=much improved; 3=minimally improved; 4=no change from baseline (the initiation of treatment); 5=minimally worse; 6= much worse; 7=very much worse since the initiation of treatment.
Time Frame: 2-month
Population: One participant did not participate in the clinicial interview.
Measure: Count of Participants; unit: Participants
Arm/Group | Active
Number analyzed (Participants) | 22
Participants
  CGI-I score of "1", "2" or "3" | 21
  CGI-I score of "4" or higher | 1

6. Secondary Outcome: Change in Behavior Rating Inventory of Executive Function (BRIEF) - Global Executive Composite - at Baseline and 2 Months Follow up
Description: The BRIEF is a standardized measure that captures views of executive functions or self-regulation in the everyday environment. The BRIEF is composed of 86 items, where each item is rated by the parent, using a 3-point Likert scale ranging from 1 ('Never') to 3 ('Often'). Total score ranges between 86 to 258. The Global Executive Composite (GEC) is an overarching summary score that incorporates all of the BRIEF clinical scales. High scores indicate executive deficit.
Time Frame: Baseline, 2-month
Population: Four participants did not complete the questionnaire.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Active
Number analyzed (Participants) | 19
score on a scale
  Baseline | 161.47 (2.97)
  End of study | 153.89 (4.13)
Statistical Analysis 1: Comparison: Active; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.035, t-test, 2 sided; Mean Difference (Final Values) = 7.58

7. Secondary Outcome: Change in Conners' Continuous Performance Test-3 (CPT-3) - Detectability (d') at Baseline and 2 Months Follow up
Description: Conners' Continuous Performance Test-3 (CPT-3) is an objective test of attention and impulsivity that has been validated in individuals aged 8 years and older.
  d-prime (d') is a measure of how well the respondent discriminates nontargets (i.e., the letter X) from targets (i.e., all other letters). This variable is also a signal detection statistic that measures the difference between the signal (targets) and noise (non-targets) distributions. In general, the greater the difference between the signal and noise distributions, the better the ability to distinguish non-targets and targets.
  CPT scores are age and gender standardized T-scores, in which the mean is equal to 50 and the standard deviation is equal to 10. d' is reverse-scored so that higher raw score and T-score values indicate worse performance (i.e., poorer discrimination). Atypical scores are higher than 60 indicating "elevated" to "very elevated" performance.
Time Frame: Baseline, 2 months
Population: One participant did not complete the test.
Measure: Mean (Standard Error); unit: T-score
Arm/Group | Active
Number analyzed (Participants) | 22
T-score
  Baseline | 50.55 (1.64)
  End of study | 51.68 (1.70)
Statistical Analysis 1: Comparison: Active; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = .521, t-test, 2 sided; Mean Difference (Final Values) = -1.13

ADVERSE EVENTS:
Time Frame: Adverse event data was collected during the two-month intervention period.
Description: No serious adverse events were reported, and no events led to intervention discontinuation. All side effects were transient, reported to be mild or moderate, and resolved after the removal of the glasses.
Arm/Group | Active
All-Cause Mortality (participants affected / at risk) | 0/24
Serious Adverse Events (participants affected / at risk) | 0/24
Other Adverse Events (participants affected / at risk) | 15/24
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Active (N=24)
Headache (General disorders) | 10
Eyestrain (General disorders) | 4
Discomfort (General disorders) | 1
Dizziness (General disorders) | 2
Tiredness (General disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-02-01): https://cdn.clinicaltrials.gov/large-docs/36/NCT05835336/Prot_SAP_000.pdf